CLINICAL TRIAL: NCT06174688
Title: A Phase 3, Multi-center, Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Safety and Efficacy of BOTOX® (Botulinum Toxin Type A) Purified Neurotoxin Complex for the Treatment of Moderate to Severe Forehead Lines in China
Brief Title: A Study to Assess the Adverse Events and Effectiveness of BOTOX Injections for the Treatment of Moderate to Severe Forehead Lines in Chinese Adult Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M22-043
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Forehead Lines
Keywords: Forehead Lines; BOTOX; Botulinum Toxin Type A
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BOTOX (Experimental): BOTOX will be injected on Day 1
  Interventions: Drug: BOTOX
- Placebo (Placebo Comparator): Placebo will be injected on Day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BOTOX — Intramuscular Injections
  Other Names: Botulinum Toxin Type A
  Arms: BOTOX
Drug: Placebo — Intramuscular Injections
  Arms: Placebo

SUMMARY:
Facial lines (such as glabellar lines [GL], lateral canthal lines [LCL], and forehead lines [FHL]) are perhaps the most visible signs of aging. Hyperfunctional facial lines that develop from repeated facial expression may be treated by selectively weakening specific muscles with small quantities of botulinum toxin. The purpose of this study is to assess adverse events and effectiveness of BOTOX in Chinese adults with moderate to severe FHL.

Participants are placed in 1 of 2 groups, called treatment arms. Around 140 adult participants with moderate to severe FHL will be enrolled in the study.

Participants in the treatment group will receive intramuscular injections on Day 1 and followed for up to 180 Days.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at the study site. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient visual acuity without the use of eyeglasses (contact lens use acceptable) to accurately assess their facial wrinkles.
* Participant must have symmetrical FHL of moderate or severe rating at maximum contraction as assessed by both investigator and participant using the Facial Wrinkle Scale with Asian Photonumeric Guide (FWS-A) at Day 1 prior to study treatment.
* Participant must have glabellar lines (GL) severity of moderate or severe rating at maximum contraction as assessed by investigator using the FWS-A at Day 1 prior to study treatment.

Exclusion Criteria:

* Participants with history of known immunization or hypersensitivity to any botulinum toxin serotype.
* Participants with history of an allergic reaction or significant sensitivity to constituents of the study drug (and its excipients) and/or other products in the same class.
* Presence of tattoos, jewelry, or clothing which obscures or interferes with the target area of interest and cannot be removed.
* Participant with history of treatments to the mid- or upper face.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who Achieved 'None' or 'Mild' on Facial Wrinkle Scale with Asian Photonumeric Guide (FWS-A) According to the Investigator Assessment of Forehead Lines (FHL) Severity | Day 30
  The investigator assesses FHL severity using the FWS-A 4-point scale ranging from 0=None to 3=Severe.
Percentage of Participants who Achieved 'None' or 'Mild' on FWS-A According to the Participant Assessment of FHL Severity | Day 30
  The participant assesses FHL severity using the FWS-A 4-point scale ranging from 0=None to 3=Severe.
Number of Participants with Adverse Events (AEs) | Day 180
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.

SECONDARY OUTCOMES:
Percentage of Participants who Achieved at least 1-Grade Improvement from Baseline on FWS-A According to the Investigator Assessment of FHL Severity | Baseline to Day 30
  The investigator assesses FHL severity using the FWS-A 4-point scale ranging from 0=None to 3=Severe.
Percentage of Participants with Responder Status of 'Very Satisfied' or 'Mostly Satisfied' on Satisfaction with Treatment on the Facial Line Satisfaction Questionnaire (FLSQ) follow up Item 5 | Day 60
  The FLSQ consists of 13 questions that assess treatment satisfaction and psychosocial impact. Participants assessed their satisfaction with FHL using the FLSQ 5-point scale ranging from -2=Very dissatisfied to 2=Very satisfied.
Percentage of Participants with Responder Status of 'Very Satisfied' or 'Mostly Satisfied' on Satisfaction with Natural Look on the FLSQ follow up Item 4 | Day 30
  The FLSQ consists of 13 questions that assess treatment satisfaction and psychosocial impact. Participants assessed their satisfaction with FHL using the FLSQ 5-point scale ranging from -2=Very dissatisfied to 2=Very satisfied.
Percentage of Participants who Achieved at Least a 20-Point Psychosocial Impact Improvement from Baseline on the FLSQ Impact Domain | Baseline to Day 30
  The FLSQ consists of 13 questions that assess treatment satisfaction and psychosocial impact. Participants assessed their satisfaction with FHL using the FLSQ 5-point scale ranging from -2=Very dissatisfied to 2=Very satisfied.
Percentage of Participants who Achieved at least 2-Grade Improvement from Baseline on FWS-A According to the Investigator Assessment of FHL Severity | Baseline to Day 30
  The investigator assesses FHL severity using the FWS-A 4-point scale ranging from 0=None to 3=Severe.
Percentage of Participants who Achieved at least 2-Grade Improvement from Baseline on FWS-A According to the Participant Assessment of FHL Severity | Baseline to Day 30
  The participant assesses FHL severity using the FWS-A 4-point scale ranging from 0=None to 3=Severe.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (12):
- China (12):
  - Beijing Hospital /ID# 250059, Beijing, Beijing Municipality
  - Peking University First Hospital /ID# 249912, Xicheng District, Beijing Municipality
  - Guangdong Second Provincial General Hospital /ID# 250742, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-Sen University /ID# 250148, Guangzhou, Guangdong
  - Peking university shenzhen hospital /ID# 249913, Shenzhen, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 250022, Wuhan, Hubei
  - Nanjing Drum Tower Hospital /ID# 250020, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University /ID# 249970, Nanjing, Jiangsu
  - Huashan Hospital, Fudan University /ID# 249854, Shanghai, Shanghai Municipality
  - Tangdu Hospital of The Fourth Military Medical University, PLA /ID# 249856, Xi’an, Shanxi
  - West China Hospital, Sichuan University /ID# 250474, Chengdu, Sichuan
  - Zhejiang Provincial People's Hospital /ID# 250120, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M22-043#additional-resources-section